CLINICAL TRIAL: NCT03107650
Title: Preoperative Prediction Model of Pathological Outcomes (Mesorectum Quality and Positive Circumferential Resection Margin) in Patients With Mid-low Rectal Cancer
Acronym: PREMARE
Status: Completed | Type: Observational
Sponsor: Pere Planellas Giné (Other)
Responsible Party: Sponsor-Investigator, Pere Planellas Giné, MD PhD, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Organization: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Other Study IDs: 0485762
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High risk patients: Patients with high risk of suboptimal mesorectum quality and/or positive circumferential margin after the application of the preoperative prediction model developed
  Interventions: Procedure: Transanal total mesorectal excision of rectal cancer
- Low risk patients: Patients with low risk of suboptimal mesorectum quality and/or positive circumferential margin after the application of the preoperative prediction model developed

INTERVENTIONS:
Procedure: Transanal total mesorectal excision of rectal cancer — To perform a total mesorectal excision through a transanal approach
  Groups: High risk patients

SUMMARY:
Elaboration of a preoperative prediction model of the quality of the mesorectum and the involvement of the circumferential margin in patients with mid-low rectal cancer who undergo laparoscopic anterior rectal resection.

In a second phase the investigators will study the utility of the prediction model in classifying patients with high risk of suboptimal quality of mesorectum and/or positive circumferential margin. Patients with high preoperative risk will undergo a transanal total mesorectal excision and patients with low risk a laparoscopic transabdominal mesorectal excision. The investigators finally will compare pathological outcomes ( quality of mesorectum and circumferential margin), survival and recurrence between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients directed to laparoscopic anterior rectal resection through a transabdominal or a transanal approach.
* Age ≥ 18 years
* Histology of adenocarcinoma or adenoma
* With or without neoadjuvant chemoradiotherapy
* TNM classification: T2 or T3, any N stage or M stage
* Intention of resection R0

Exclusion Criteria:

* TNM classification: T1 or T4.
* Complicated rectal cancer or emergency surgery.
* Previous major colorectal surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected of mid-low rectal cancer
Sampling Method: Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the quality of mesorectum in the rectal specimen according to international consensus (goog quality, moderate quality and poor quality) | 30 days
  Evaluation of the quality of mesorectum as optimal or suboptimal (international consensus defines three grades of resection:
  Group 1: including mesorectal resection, good quality Group 2: intramesorectal resection: moderate quality Group 3: resection in the muscularis propria, poor quality).
  Investigators will group patients into two groups: optimal mesorectum (group 1) and suboptimal mesorectum (group 2-3).
Evaluation of the circumferential margin status in the rectal specimen according international consensus (positive margin if tumor ≤ 1mm from circumferential margin) | 30 days
  Evaluation of the circumferential margin status (positive or negative) in the rectal specimen according international consensus (positive margin if tumor ≤ 1mm from circumferential margin)

SECONDARY OUTCOMES:
Recurrence | 2 years
  Rate of tumor recurrence
Survival | 2 years
  Rate of survival

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Dr. Josep Trueta of Girona, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Planellas P, Marinello F, Elorza G, Golda T, Farres R, Espin-Basany E, Enriquez-Navascues JM, Kreisler E, Cornejo L, Codina-Cazador A. Extended Versus Standard Complete Mesocolon Excision in Sigmoid Colon Cancer: A Multicenter Randomized Controlled Trial. Ann Surg. 2022 Feb 1;275(2):271-280. doi: 10.1097/SLA.0000000000005161. PMID 34417367
- [Derived] Planellas P, Salvador H, Cornejo L, Buxo M, Farres R, Molina X, Maroto A, Ortega N, Rodriguez-Hermosa JI, Codina-Cazador A. Risk factors for suboptimal laparoscopic surgery in rectal cancer patients. Langenbecks Arch Surg. 2021 Mar;406(2):309-318. doi: 10.1007/s00423-020-02029-0. Epub 2020 Nov 27. PMID 33244719